CLINICAL TRIAL: NCT05315466
Title: Comparison Between Surgical and Conservative Treatment for Lumbar Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF MINSAL2009.STENOSI
Record Dates: First submitted 2017-03-01; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2017-03

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients affected by lumbar spinal stenosis who are designated to surgical or conservative treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical treatment (Experimental): Different types of non-surgical treatments
  Interventions: Procedure: Non-surgical treatment
- Surgical treatment (Experimental): Surgical treatment for spinal stenosis
  Interventions: Procedure: Surgical treatment for spinal stenosis

INTERVENTIONS:
Procedure: Non-surgical treatment — Analgesics, anti-inflammatories, muscle relaxants, physical therapy, Global Postural Rehabilitation, magnetic therapy, laser therapy, transcutaneous electrical nervous stimulation (TENS), massage, cognitive-behavioral therapy and all those procedures that can bring benefit to back and leg pain.
  Arms: Non-surgical treatment
Procedure: Surgical treatment for spinal stenosis — Decompression of nerve structures by laminotomy or laminectomy and posterior lumbar fusion if stabilization of the column is required.
  Arms: Surgical treatment

SUMMARY:
This study aims to compare the outcomes of surgical treatment and conservative treatment at medium- and long-term period (minimum 2 years) in patients with lumbar stenosis who come to the observation of the PI's Team at the Rizzoli Orthopaedic Institute, through a series exhaustive questionnaires to self-administer to patients in order to define a path of "decision-making" as effective as possible for the patient and the doctor.

DETAILED DESCRIPTION:
Non-surgical treatment:

Conservative treatment may include different approaches, such as analgesics, anti-inflammatories, muscle relaxants, physical therapy, Global Postural Rehabilitation, magnetic therapy, laser therapy, TENS, massage, cognitive-behavioral therapy and all those procedures that can bring benefit in back and legs pain.

Surgical treatment:

Surgical treatment of lumbar stenosis is the decompression surgery which relieves the nerve structures to prevent permanent neurological damage. Decompression can be made on one or more segments of the spine and can be done with laminectomy, hemilaminectomy, laminotomy.

During a laminotomy part of the vertebral lamina is removed above and below the compressed nerve. The opening created is sometimes enough to relieve the compression on the nerve. In most cases, also the disc material and bone spur that compress the nerve are removed.

During a laminectomy the vertebral lamina is completely removed, along with the disc and the bone material that compress the nerves. The opening produced by the removal of the lamina is protected by back muscles and ligaments.

If the damage has occurred at several levels and bone of the vertebral support structures must be removed to achieve decompression, it can be performed a stabilization surgery with vertebral bone fusion (arthrodesis) in order to avoid instability of the column. Fusion is carried out to eliminate the mobility between different vertebrae and it is achieved using bone derived from the patient's iliac crest or from a donor. The bone gradually grows and melts with the same vertebrae. This limits the movements that may have been one of the causes of back pain. It takes about six months for it to achieve a solid bony spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmatory imaging study (MRI or CT) showing lumbar spinal stenosis at one or more levels (L2 to sacrum) defined as narrowing of the central spinal canal, lateral recesses, or neural foramens due to encroachment on the neural structures by the surrounding bone and soft tissue.

Exclusion Criteria:

* Patients are not eligible if they have evidence of instability on lateral flexion- extension radiographs, defined as a change of #10° of angulation of adjacent segments by Cobb measurement or a change of more than 4 mm of anteroposterior or posteroanterior translation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08-08 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Back and leg pain assessed by VAS | Change from baseline VAS at 3, 6, 12, 24 months
  Self-administered questionnaires for patients to evaluate back and leg pain (VAS score)
Functional activity assessed by ODI | Change from baseline ODI at 3, 6, 12, 24 months
  Self-administered questionnaires for patients to evaluate a disability index (ODI)
Quality of life assessed by EQ-5D | Change from baseline EQ-5D at 3, 6, 12, 24 months
  Self-administered questionnaires for patients to evaluate the quality of life (EQ-5D)

SECONDARY OUTCOMES:
Complications | 6, 12, 24 months
  Evaluation of complications associated to the surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gasbarrini, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacs FM, Urrutia G, Alarcon JD. Surgery versus conservative treatment for symptomatic lumbar spinal stenosis: a systematic review of randomized controlled trials. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1335-51. doi: 10.1097/BRS.0b013e31820c97b1. PMID 21311394
- [Background] Amundsen T, Weber H, Nordal HJ, Magnaes B, Abdelnoor M, Lilleas F. Lumbar spinal stenosis: conservative or surgical management?: A prospective 10-year study. Spine (Phila Pa 1976). 2000 Jun 1;25(11):1424-35; discussion 1435-6. doi: 10.1097/00007632-200006010-00016. PMID 10828926
- [Background] Malmivaara A, Slatis P, Heliovaara M, Sainio P, Kinnunen H, Kankare J, Dalin-Hirvonen N, Seitsalo S, Herno A, Kortekangas P, Niinimaki T, Ronty H, Tallroth K, Turunen V, Knekt P, Harkanen T, Hurri H; Finnish Lumbar Spinal Research Group. Surgical or nonoperative treatment for lumbar spinal stenosis? A randomized controlled trial. Spine (Phila Pa 1976). 2007 Jan 1;32(1):1-8. doi: 10.1097/01.brs.0000251014.81875.6d. PMID 17202885
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Blood E, Hanscom B, Herkowitz H, Cammisa F, Albert T, Boden SD, Hilibrand A, Goldberg H, Berven S, An H; SPORT Investigators. Surgical versus nonsurgical therapy for lumbar spinal stenosis. N Engl J Med. 2008 Feb 21;358(8):794-810. doi: 10.1056/NEJMoa0707136. PMID 18287602
- [Background] Zucherman JF, Hsu KY, Hartjen CA, Mehalic TF, Implicito DA, Martin MJ, Johnson DR 2nd, Skidmore GA, Vessa PP, Dwyer JW, Puccio ST, Cauthen JC, Ozuna RM. A multicenter, prospective, randomized trial evaluating the X STOP interspinous process decompression system for the treatment of neurogenic intermittent claudication: two-year follow-up results. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1351-8. doi: 10.1097/01.brs.0000166618.42749.d1. PMID 15959362